CLINICAL TRIAL: NCT00946426
Title: Insulin Resistance in Type I Diabetes in Pediatric Care
Status: Withdrawn | Type: Observational
Why Stopped: PI left institution
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Dana S. Hardin, The Research Institute at Nationwide Children's Hospital
Other Study IDs: IRB09-00160
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Constriction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic: Hyperinsulinemic euglycemic clamp
  Interventions: Other: Clamp

INTERVENTIONS:
Other: Clamp — Insulin sensitivity, Hepatic glucose production, Evaluation of inflammation, Socioeconomic status, Ethnicity and family history

SUMMARY:
24 children (12 African-American, Hispanic, or American Indian, 12 Caucasian) previously diagnosed with type 1 diabetes mellitus will participate in this pilot study to evaluate the presence of hepatic and peripheral insulin resistance. The investigators will use this pilot information to test the hypothesis that insulin resistance occurs in some children with type 1 DM, is secondary to underlying risk factors, and is responsible for increased insulin needs. Methods will include a "step-up" hyperinsulinemic euglycemic clamp and infusion of the stable isotope 6,6-[2H2]-glucose. Patient and parent interviews will be conducted to gather information about nutritional intake, ethnicity, family history, and socioeconomic status. The investigators will also measure inflammatory cytokines and free fatty acids to determine whether they are associated with differences in insulin resistance among type 1 diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with type 1 diabetes
* ages 9 -11 tanner 1 or 16-23 tanner 4-5

Exclusion Criteria:

* None

Ages: 9 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Endocrinology clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline

SECONDARY OUTCOMES:
Hepatic glucose output | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dana S Hardin, MD, Principal Investigator — The Research Institute at Nationwide Children's Hospital, The Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States